CLINICAL TRIAL: NCT07234058
Title: A Non-Comparative Phase IIR Trial Assessing Fianlimab Plus Cemiplimab Plus Pemetrexed-Platinum Chemotherapy or Cemiplimab Plus Pemetrexed-Platinum Chemotherapy for Treatment-Naive Pleural Mesothelioma (PM) Patients
Brief Title: Trial Assessing Fianlimab Plus Cemiplimab Plus Chemotherapy or Cemiplimab Plus Chemotherapy in Patients With Pleural Mesothelioma
Acronym: LAG-MAPS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-2402
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pleural Mesotheliomas
Keywords: pleural mesothelioma; cemiplimab; fianlimab; anti-LAG3; anti-PD-1
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — cemiplimab; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Intervention Model Description: The parallel arms are not comparative.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: cemplimab + chemotherapy (Other): cemplimab 350mg administered every 3 weeks for up to 24 months, with pemetrexed 500 mg/m² + platinum salt (cisplatin 75 mg/m² or carboplatin AUC 5) for 6 cycles of 21 days.
  Interventions: Drug: Cemiplimab; Drug: Pemetrexed (Alimta); Drug: Cisplatin; Drug: Carboplatin (AUC 5)
- Arm B: cemplimab + fianlimab + chemotherapy (Experimental): cemplimab 350mg and fianlimab 1600mg administered every 3 weeks for up to 24 months, with pemetrexed 500 mg/m² + platinum salt (cisplatin 75 mg/m² or carboplatin AUC 5) for 6 cycles of 21 days.
  Interventions: Drug: Cemiplimab; Drug: Fianlimab; Drug: Pemetrexed (Alimta); Drug: Cisplatin; Drug: Carboplatin (AUC 5)

INTERVENTIONS:
Drug: Cemiplimab — 350mg every 3 weeks for up to 24 months.
  Other Names: Libtayo
Drug: Fianlimab — 1600mg every 3 weeks for up to 24 months.
  Arms: Arm B: cemplimab + fianlimab + chemotherapy
Drug: Pemetrexed (Alimta) — 500 mg/m² every 3 weeks for 6 cycles.
  Other Names: Alimta
Drug: Cisplatin — 75 mg/m² every 3 weeks for 6 cycles.
Drug: Carboplatin (AUC 5) — AUC 5 (recommended maximum dose of 800 mg) every 3 weeks for 6 cycles.

SUMMARY:
This is a multicentre, phase IIR, double non-comparative arm trial, with an initial safety run for the anti-LAG3 arm.

Approximately 40 sites will participate in the study and will enroll 126 patients with treatment-naive, unresectable malignant PM.

Treatment will be administered in 21-day cycles and will continue until disease progression, unacceptable toxicity, withdrawal of consent or for 2 years immunotherapy maximum.

Once the patient discontinues study treatment, the treatment period will end and the patient will enter the follow-up period. No cross-over is allowed between arms.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written Informed Consent.

   * Subjects must have signed and dated an IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal subject care.
   * Subjects must be willing and able to comply with scheduled visits, treatment schedule, and laboratory testing.
2. Histological diagnosis (no cytology allowed, thoracoscopy biopsy recommended).
3. Non resectable PM as evaluated by a specialist MTB comprising a specialized thoracic surgeon.
4. Measurable disease by CT with iodure injection according to RECIST 1.1 modified criteria for mesothelioma (pleural thickness perpendicular to the chest wall or mediastinum of 7 mm or more, on 2 positions, at 3 separate levels on transverse cuts of CT-scan, at least 1 cm apart, the sum of 6 measurements defining a pleural unidimensional measure), or according to RECIST1.1 criteria for mediastinal nodes or metastatic lesion.
5. ECOG PS 0 and 1.
6. Weight loss <10% within 3 months of study entry.
7. Chemo-naive and immuno-naive.
8. Age ≥18 years, <76 years.
9. Life expectancy >3 months.
10. Available pathological samples (at least 10 slides from the thoracoscopy pleural biopsy sample).
11. Adequate biological functions: creatinine clearance ≥45 mL/min (Cockroft or MDRD or CKD-epi); neutrophils ≥1500/mm3; platelets ≥100 000/mm3; haemoglobin ≥9g/dL; AST and ALT <3 x ULN, total bilirubin <2 x ULN (patients with hepatic metastases or Gilbert's syndrome must have AST and ALT ≤5 x ULN and a baseline total bilirubin ≤2 x ULN).
12. WOCBP* must have a negative serum (beta-hCG) at screening.

    *WOCBP are defined as women who are fertile following menarche until becoming postmenopausal, unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high FSH level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient to determine the occurrence of a postmenopausal state. The above definitions are according to the CTFG guidance. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.
13. Male study participants with WOCBP partners are required to use condoms during the study and until 6 months after the last dose of study treatment unless they are vasectomised or practice sexual abstinence.
14. Vasectomised partner or vasectomised study participant must have received medical assessment of the surgical success.

    NB: Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and LAM are not acceptable methods of contraception. Female condom and male condom should not be used together.
15. WOCBP must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the entire trial and until 6 months after last treatment.
16. All men must agree not to donate sperm during the trial and for 6 months after receiving the last therapy dose.
17. As recommended in current French guidelines, a firm recommendation of radiation therapy for thoracocentesis tracts (3 x 7Gy) is made for patients with thoracocentesis or thoracoscopy within 2 months before accrual, with a firmly recommended interval between thoracoscopic procedure (removal of drains) and radiation of no more than 42 days. A 7-day interval between the end of radiotherapy and the initiation of treatment should be respected.

Exclusion Criteria:

1. ECOG PS>2.
2. Previous cancer treatment including chemotherapy or immunotherapy with anti-PD-1, anti-PD-L1, Anti-CTLA4 or any ICI antibody.
3. Pleural effusion as the only radiological abnormality without measurable pleural thickness or mediastinal node enlargement.
4. Peritoneal, pericardial or tunica vaginalis testis mesothelioma.
5. Previous diagnosis of adenocarcinoma from any anatomic site within the previous 5 years, with the exception of prostate adenocarcinoma history within the previous 5 years, in case of localized prostate cancer, with good prognostic factors according to d'Amico classification (<T2a, score de Gleason ≤6 and PSA ≤10 ng/ml) provided they were treated in a curative way (surgery or radiotherapy, without any chemotherapy). Previous or active cancer within the previous 5 years (except for treated carcinoma in situ of the cervix, or basal cell skin cancer treated or not).
6. Uncontrolled pleural effusion requiring frequent thoracocentesis (needing thoracoscopic pleural pleurodesis before possible accrual).
7. Symptomatic untreated brain metastasis (without previous whole brain radiotherapy or stereotactic ablative brain radiotherapy or without surgical resection). At least 2 weeks delay between the end of radiotherapy and the beginning of immuno-chemotherapy treatment should be respected. Asymptomatic brain metastasis, not needing corticosteroids greater than 10 mg prednisone equivalent daily or mannitol infusions, are allowed.
8. Radiotherapy needed at initiation of tumour treatment, except bone palliative radiotherapy on a painful or compressive metastasis, or radiotherapy on thoracic drain or puncture routes.
9. History of previous primary immunodeficiency, organ transplantation needing an immunosuppressive treatment, any immunosuppressive drug within 28 days before randomisation date, or history of severe toxicity (grade 3/4) by immune mechanism linked to another immunotherapy treatment for any kind of disease.
10. Systemic treatment with corticosteroids with greater dose than 10 mg prednisone equivalent daily, within 14 days before initiation of the treatment. Inhaled, nasal or topic corticosteroids are allowed.
11. History of active autoimmune disease, needing systemic immunosuppressive drug, including but not limited to rheumatoid polyarthritis, myasthenia, autoimmune hepatitis, systemic Lupus, Wegener's granulomatosis, vascular thrombosis associated with anti-phospholipid syndrome, Sjogren's syndrome with interstitial pulmonary disease, recent Guillain-Barré syndrome within previous 15 years, multiple sclerosis, vasculitis, or glomerulonephritis.

    Patients with type I diabetes, or hypothyroidy, or immune cutaneous disease (vitiligo, psoriasis, alopecia) or benign rheumatoid polyarthritis not needing any immunosuppressive systemic treatment or over 10 mg daily oral steroids, or benign sicca syndrome (Sjogren) without interstitial pulmonary disease, or history of past Guillain-Barré syndrome beyond 15 previous years, totally reversible with no sequalae, no systemic immunosuppressive treatment during the last 20 years, can be included. Patients with Grave's disease or psoriasis not requiring systemic therapy within the last two years from randomisation can be included.
12. Active inflammatory intestinal disease (diverticulosis, Crohn disease, haemorrhagic recto-colitis, coeliac disease) requiring systemic treatment, or any serious chronic intestinal disease with uncontrolled diarrhoea.
13. History or current evidence of significant (CTCAE grade ≥2) local or systemic infection (e.g. cellulitis, pneumonia, septicaemia) requiring systemic antibiotic treatment within 2 weeks prior to the first dose of trial medication.
14. Active uncontrolled infection requiring therapy including active tuberculosis. Past primary pulmonary tuberculosis in youth does not consist of a contra-indication. Past tuberculosis disease history does not consist of a contra-indication provided the patient was treated during at least 6 months by anti-tuberculosis antibiotic treatment.
15. Uncontrolled infection with HIV, HBV, or HCV infection; or diagnosis of immunodeficiency that is related to, or results in chronic infection.

    Notes:
    1. Patients with known HIV who have controlled infection (undetectable viral load and CD4 count above 350 either spontaneously or on a stable antiviral regimen) are permitted. For patients with controlled HIV infection, monitoring will be performed per local standards.
    2. Patients with known hepatitis B (HepBsAg+) who have controlled infection (serum hepatitis B virus DNA PCR that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) are permitted. Patients with controlled infections must undergo periodic monitoring of HBV DNA per local standards and must remain on anti-viral therapy for at least 6 months beyond the last dose of investigational study drug.
    3. Patients who are known hepatitis C virus antibody positive (HCV Ab+) who have controlled infection (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted.
    4. Patients with HIV or hepatitis must be reviewed by a qualified specialist (e.g. infectious disease or hepatologist) managing this disease prior to commencing and regularly throughout the duration of their participation in the trial.
16. Received a live vaccine within 30 days of planned start of study medication. Live or live attenuated vaccination with replicating potential. If a patient intends to receive a COVID-19 vaccine before the start of study drug, participation in the study should be delayed at least 1 week after any COVID-19 vaccination. During the treatment period, it is recommended to delay COVID-19 vaccination until patients are receiving and tolerating a steady dose of study drug. A vaccine dose should not be less than 48 hours before or after study drug dosing. mRNA and adenovirus vector anti-SARS-CoV2 vaccine are allowed.
17. General serious condition such as congestive uncontrolled cardiac failure, uncontrolled cardiac arrythmia, uncontrolled ischemic cardiac disease (unstable angina or history of myocardial infarction within the previous 6 months), history of stroke within the 6 previous months, history of myocarditis. Patients with a significant cardiac history, even if controlled, should have a LVEF >45%.
18. TnT or troponin I TnI > 2x institutional ULN at baseline. Patients with TnT or TnI levels between >1 to 2xULN are permitted if repeat levels within 24 hours are ≤ 1x ULN. If TnT or TnI levels are >1 to 2xULN within 24 hours, the subject may undergo a cardiac evaluation and be considered for treatment by the investigator based on cardiological medical judgement in the patient's best interest.
19. Known hypersensitivity to the active substances or to any of the excipients.
20. Pre-existing moderate or severe lung interstitial disease as assessed by the diagnosis CT-scan and decrease of TLCO higher than 35% from theoretical normal values linked to such interstitial disease.
21. Inability to comply with study or follow-up procedures as estimated by the referent investigator.
22. Pregnant or breastfeeding women.
23. Women of childbearing potential (WOCBP)* who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 6 months after the last dose. Highly effective contraceptive measures include:

    1. Stable use of combined (oestrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation initiated 2 or more menstrual cycles prior to screening;
    2. Intrauterine device; intrauterine hormone-releasing system;
    3. Bilateral tubal occlusion/ligation;
    4. Vasectomized partner (provided that the male vasectomized partner is the sole sexual partner of the WOCBP study participant and that the vasectomized partner has obtained medical assessment of surgical success for the procedure); or
    5. Sexual abstinence†. *Pregnancy testing and contraception are required for WOCBP. †Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drugs. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.
24. For patients receiving cisplatin: patients with hearing problems; creatinine clearance <60 ml/min; patients concomitantly receiving phenytoin with prophylactic aim.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the activity of the combination of double immunotherapy anti-LAG3+ anti-PD-1 and pemetrexed+platinum chemotherapy | 6 months after randomisation.
  The primary endpoint is 6-month disease control rate (DCR). The analysis will be conducted in the FAS population. DCR is defined as the proportion of patients who have achieved at 6 months an overall response of CR, PR or stable disease (SD), as assessed by an independant review committee (IRC) per RECIST v1.1 modified for mesothelioma.

SECONDARY OUTCOMES:
Tolerance, safety of treatment | From time of informed consent through treatment period and up to 90 days post last dose of study treatment (maximum of 2 years and 3 months).
  Incidence, nature, and severity of adverse events (AE), graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0). The rate of Hyper-Progressive Disease (HPD) will also be calculated.
Progression Free Survival (PFS) as assessed by an IRC | At progression, up to 2 years after start of treatment.
  PFS is defined as the time between the date of randomisation and the first date of documented progression, as assessed by investigator and an IRC per RECIST v1.1 modified for mesothelioma, or death due to any cause, whichever occurs first.
PFS as assessed by the investigator | At progression, up to 2 years after start of treatment.
  PFS is defined as the time between the date of randomisation and the first date of documented progression, as assessed by investigator and an IRC per RECIST v1.1 modified for mesothelioma, or death due to any cause, whichever occurs first.
PFS according to the histological subtype epithelioid vs. non-epithelioid | At progression, up to 2 years after start of treatment.
  PFS is defined as the time between the date of randomisation and the first date of documented progression, as assessed by investigator and an IRC per RECIST v1.1 modified for mesothelioma, or death due to any cause, whichever occurs first. PFS will be analysed according to the histological subtype.
Overall Survival (OS) | Around 42 months.
  OS is defined as the time from date of randomisation to the date of death due to any cause. If a death has not been observed by the date of the analysis cut-off, OS will be censored at the date of last contact.
Best Overall Response Rate (ORR) | At progression, up to 2 years after start of treatment.
  ORR is defined as the proportion of patients who have achieved a best overall response of complete response (CR) or partial response (PR) as determined by investigator review of radiographic disease assessments per RECIST v1.1 modified for mesothelioma.
Time until definitive HRQol score deterioration | At progression, up to 2 years after start of treatment.
  Time until definitive HRQol score deterioration will be measured using LCSS-meso questionnaire.
General health status | At progression, up to 2 years after start of treatment.
  General health status will be measured using the EQ-5D-5L questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Myriam LOCATELLI-SANCHEZ, Principal Investigator — Hôpital Lyon-Sud, Hospices Civils de Lyon; Pr Gérard ZALCMAN, Principal Investigator — Hôpital Bichat, AP-HP
Locations (37):
- France (37):
  - Aix-Pertuis - CHI, Aix-en-Provence
  - Amiens - CHU, Amiens
  - Angers - CHU, Angers
  - Avignon - CH, Avignon
  - Besançon - CHU, Besançon
  - Bordeaux - Institut Bergonié, Bordeaux
  - Boulogne - APHP Ambroise Paré, Boulogne-Billancourt
  - Caen - CHU, Caen
  - Clermont-Ferrand - Centre Jean Perrin, Clermont-Ferrand
  - Clermont-Ferrand - CHU, Clermont-Ferrand
  - Créteil - CHI, Créteil
  - Dijon - Centre Georges-François Leclerc, Dijon
  - Grenoble - CHU, Grenoble
  - La Roche-Sur-Yon - CHD Vendée, La Roche-sur-Yon
  - Le Mans - CHG, Le Mans
  - Lille - CHU, Lille
  - Marseille - APHM Nord, Marseille
  - Marseille - Hôpital Européen, Marseille
  - Montpellier - CHU, Montpellier
  - Mulhouse - GHRMSA, Mulhouse
  - Nantes - Hôpital Laennec, Nantes
  - Paris - APHP Bichat, Paris
  - Paris - APHP Cochin, Paris
  - Bordeaux - CHU, Pessac
  - Lyon - HCL, Pierre-Bénite
  - Reims - Institut Godinot, Reims
  - Rennes - CHU, Rennes
  - Nantes - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Saint-Nazaire - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - Toulon - CHI, Toulon
  - Toulon - Sainte Anne HIA, Toulon
  - Toulouse - CHU, Toulouse
  - Tours - CHU, Tours
  - Vandoeuvre-lès-Nancy - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Villefranche sur Saône - CH, Villefranche-sur-Saône
  - Villejuif - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data underlying the results reported in this article, as well as the study protocol and statistical analysis plan, will be made available after deidentification immediately following publication and for three years. Researchers who provide a methodologically sound proposal for any purpose may direct proposals to contact@ifct.fr. To gain access, data requestors will need to sign a data access agreement that requires approval by the French Cooperative Thoracic Intergroup.

REFERENCES:
- See also: IFCT website — https://www.ifct.fr/